CLINICAL TRIAL: NCT05020600
Title: Investigation of the Effect of Initial Central Sensitization Severity on Treatment Response in Patients With Fibromyalgia
Brief Title: The Effect of Central Sensitization on Treatment Response in Patients With Fibromyalgia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: 09.2021.117
Record Dates: First submitted 2021-08-18; First posted 2021-08-25 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2022-11

CONDITIONS: Central Sensitisation; Fibromyalgia
MeSH Terms: conditions — Fibromyalgia | interventions — Duloxetine Hydrochloride; Pregabalin; Amitriptyline

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with fibromyalgia: Patients diagnosed with fibromyalgia according to American College of Rheumatology 2016 criteria
  Interventions: Drug: Duloxetine; Drug: Pregabalin; Drug: Amitriptyline

INTERVENTIONS:
Drug: Duloxetine — First-line fibromyalgia treatment
  Other Names: Dyloxia
Drug: Pregabalin — First-line fibromyalgia treatment
  Other Names: Lyrica
Drug: Amitriptyline — First-line fibromyalgia treatment
  Other Names: Laroxyl

SUMMARY:
Central sensitization (CS) is as increased response to normal or sub-threshold stimuli of central nervous system and its close relationship with fibromyalgia has been demonstrated in several studies. However, the effect of initial CS severity on treatment response in these patients is not fully known. In this study, it was aimed to investigate the severity of CS and its effect on treatment response in patients with fibromyalgia.

DETAILED DESCRIPTION:
Fibromyalgia is a disease characterized by chronic widespread pain and its etiology and pathophysiology are still unknown.It is considered to be the main member of the central sensitization-related disease group known as central sensitivity syndromes with impaired pain regulation.In various studies, hyperalgesia and allodynia, which are accepted as objective findings of central sensitization in patients with fibromyalgia, strengthen the relationship between fibromyalgia and central sensitization. The central sensitization inventory (CSI) was developed in 2012 to be used in the recognition of central sensitivity syndromes in patients with fibromyalgia. A score of 40 and above is accepted in favor of central sensitization in the scale, which consists of two parts, in which central sensitization-related symptoms and diagnoses are questioned; scores of 30-39 are classified as mild, 40-49 moderate, 50-59 severe, and 60-100 very severe. Parallel to the increase in the CSI score, an increase is observed in patients' pain severity, disability, depressive symptoms and sleep disorders.In addition, it has been reported in the literature that factors such as pre-treatment pain severity and depression affect the treatment response.Considering all these factors, it is possible that there is a relationship between the severity of central sensitization and treatment response in patients with fibromyalgia.Based on this, in this study, it was aimed to investigate the effect of central sensitization severity, which was evaluated with CSI before treatment, on the treatment process.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosing fibromyalgia according to ACR 2016 criteria
* Between the ages of 18-65
* Agree to participate in the study

Exclusion Criteria:

* History of concomitant systemic inflammatory disease, active infection and malignancy
* Refusing to participate in the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Fibromyalgia patients
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-08-19 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Visual analog scale ( VAS) pain | 2 year
  Pain rating scale. The VAS consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be')
Symptom severity scale | 2 year
  The SS scale quantifies symptom severity on a 0-12 scale by scoring problems with fatigue, cognitive dysfunction and unrefreshed sleep over the past week
Fibromyalgia impact scale | 2 year
  The questionnaire was developed to determine the degree of being affected by the disease in patients with a diagnosis of fibromyalgia.The scale consists of 10 parts in total, and the first part is a Likert scale containing 11 questions. High scores indicate that the patient is overly affected.
Short Form-36 | 2 year
  Standardized questionnaire to investigate the quality of life in patients. The score of the scale is between 0-100. The higher scores are associated with greater deterioration in quality of life.
Central sensitization inventory | 2 year
  Standardized questionnaire to determine the level of central sensitization. Patients with a score of 40 and above are considered to have central sensitization.

CONTACTS AND LOCATIONS:
Overall Officials: Canan SANAL TOPRAK, assoc. prof., Study Director — Marmara University
Locations (1):
- Feyza Nur YUCEL, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Result] Woolf CJ, Thompson SW, King AE. Prolonged primary afferent induced alterations in dorsal horn neurones, an intracellular analysis in vivo and in vitro. J Physiol (Paris). 1988-1989;83(3):255-66. PMID 3272296
- [Result] Akinci A, Al Shaker M, Chang MH, Cheung CW, Danilov A, Jose Duenas H, Kim YC, Guillen R, Tassanawipas W, Treuer T, Wang Y. Predictive factors and clinical biomarkers for treatment in patients with chronic pain caused by osteoarthritis with a central sensitisation component. Int J Clin Pract. 2016 Jan;70(1):31-44. doi: 10.1111/ijcp.12749. Epub 2015 Nov 11. PMID 26558538
- [Result] Bhargava J, Goldin J. Fibromyalgia. 2025 Jan 31. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK540974/ PMID 31082018
- [Result] Pomares FB, Funck T, Feier NA, Roy S, Daigle-Martel A, Ceko M, Narayanan S, Araujo D, Thiel A, Stikov N, Fitzcharles MA, Schweinhardt P. Histological Underpinnings of Grey Matter Changes in Fibromyalgia Investigated Using Multimodal Brain Imaging. J Neurosci. 2017 Feb 1;37(5):1090-1101. doi: 10.1523/JNEUROSCI.2619-16.2016. Epub 2016 Dec 16. PMID 27986927
- [Result] Mayer TG, Neblett R, Cohen H, Howard KJ, Choi YH, Williams MJ, Perez Y, Gatchel RJ. The development and psychometric validation of the central sensitization inventory. Pain Pract. 2012 Apr;12(4):276-85. doi: 10.1111/j.1533-2500.2011.00493.x. Epub 2011 Sep 27. PMID 21951710
- [Result] Neblett R, Hartzell MM, Mayer TG, Cohen H, Gatchel RJ. Establishing Clinically Relevant Severity Levels for the Central Sensitization Inventory. Pain Pract. 2017 Feb;17(2):166-175. doi: 10.1111/papr.12440. Epub 2016 Mar 15. PMID 26989894
- [Result] Wolfe F, Clauw DJ, Fitzcharles MA, Goldenberg DL, Hauser W, Katz RL, Mease PJ, Russell AS, Russell IJ, Walitt B. 2016 Revisions to the 2010/2011 fibromyalgia diagnostic criteria. Semin Arthritis Rheum. 2016 Dec;46(3):319-329. doi: 10.1016/j.semarthrit.2016.08.012. Epub 2016 Aug 30. PMID 27916278
- See also: symptom severity (SS) scale in the diagnostic criteria for fibromyalgia — https://www.medscape.com/answers/329838-18860/what-is-the-symptom-severity-ss-scale-in-the-diagnostic-criteria-for-fibromyalgia